CLINICAL TRIAL: NCT03999892
Title: ACHIEVE-D Pilot Study
Brief Title: Adapted ACHIEVE Curriculum for Community Mental Health Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00194122; P50MH115842 (NIH)
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Results first posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Mental Disorders, Severe
MeSH Terms: conditions — Obesity; Mental Disorders | interventions — Achieve no-mix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot weight management module (Experimental): Consumers with serious mental illness who attend a psychiatric rehabilitation program will participate in a pilot of modules of a group-based diet and physical activity program. Staff/ peer leaders a psychiatric rehabilitation program will observe sessions.
  Interventions: Behavioral: ACHIEVE

INTERVENTIONS:
Behavioral: ACHIEVE — The investigators will test two modules of the adapted video-assisted curriculum format of 45 to 60-minute multipurpose classes, which will include a segment on group weight management (~20-30 minutes) and group exercise (~20-30 minutes). Within each module, the group weight management topic varies by week, and within each week the content of the three weight management groups builds gradually and is purposely repeated. Within each module, the group exercise classes will focus on mild to moderate intensity aerobic exercise using an exercise video. In this pilot study, a trained study interventionist will deliver the ACHIEVE-D curriculum.

SUMMARY:
In light of the obesity epidemic in persons with serious mental illness (SMI), there is an urgent need to scale-up behavioral interventions that have demonstrated efficacy in the clinical trial setting such as the intervention in the National Institute of Mental Health (NIMH)-funded Achieving Healthy Lifestyles in Psychiatric Rehabilitation (ACHIEVE) trial. To increase ease of adoption and sustained implementation of ACHIEVE in community mental health programs, the format needs to be adapted for delivery by community mental health staff. Based on the investigators' experience conducting the ACHIEVE trial, this study team had modified the ACHIEVE intervention into a new ACHIEVE curriculum appropriate for community mental health settings. Therefore, the investigators will pilot test 8 weeks of this curriculum in a community-based psychiatric rehabilitation program (PRP) to determine whether this format is acceptable to participating PRP consumers with SMI as well as PRP staff and peer leaders.

DETAILED DESCRIPTION:
Prevalence of obesity is significantly elevated and a leading cause of preventable death in people with serious mental illness (SMI) through its effects on other cardiovascular disease (CVD) risk factors and CVD. Behavioral interventions targeting changes in diet and exercise need to be tailored to the needs of people with SMI, such as memory impairment and limited executive function. The NIMH-funded Achieving Healthy Lifestyles in Psychiatric Rehabilitation (ACHIEVE) trial tested a behavioral weight-loss intervention for persons with SMI and demonstrated clinically significant weight loss. In light of the obesity epidemic in persons with SMI, there is an urgent need to scale-up interventions like ACHIEVE. To increase ease of adoption and sustained implementation of ACHIEVE in community mental health programs, the format needs to be adapted for delivery by community mental health staff. Based on the investigators' experience conducting the ACHIEVE trial, this study team had modified the ACHIEVE intervention into a new ACHIEVE curriculum appropriate for community mental health settings. Therefore, the investigators will pilot test 8 weeks of this curriculum in a community-based psychiatric rehabilitation program (PRP) to determine whether this format is acceptable to participating PRP consumers with SMI as well as PRP staff and peer leaders.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older
* consumers at Prologue psychiatric rehabilitation program
* expected to be in the rehabilitation program for at least 6 months after enrollment
* able to attend the intervention classes 3 days per week
* able and willing to give informed consent and participate in the intervention
* have a body mass index (BMI) over 25 kg/m2
* be interested in losing weight

Exclusion Criteria:

* any underlying medical conditions that could seriously reduce life expectancy, ability to participate in the study, or for which dietary change or physical activity may be contraindicated and/or require medical supervision by a physician (e.g., medication-dependent diabetes mellitus, cancer or malignant tumor, lung disease requiring supplemental oxygen, dementia or cognitive impairment, consumption of more than 14 drinks per week, eating disorders, angina, or diagnosis in the last 12 months of myocardial infarction, congestive heart failure, transient ischemic attack or stroke, liver disease or kidney disease)
* women who are pregnant or breastfeeding
* individuals with an inability to walk to participate in exercise class as demonstrated by walking up and down 2 flights of stairs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Daumit, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daumit GL, Dickerson FB, Wang NY, Dalcin A, Jerome GJ, Anderson CA, Young DR, Frick KD, Yu A, Gennusa JV 3rd, Oefinger M, Crum RM, Charleston J, Casagrande SS, Guallar E, Goldberg RW, Campbell LM, Appel LJ. A behavioral weight-loss intervention in persons with serious mental illness. N Engl J Med. 2013 Apr 25;368(17):1594-602. doi: 10.1056/NEJMoa1214530. Epub 2013 Mar 21. PMID 23517118

RESULTS

PARTICIPANT FLOW:
Groups:
- Consumers With SMI: Consumers with serious mental illness who attend a psychiatric rehabilitation program (PRP) will participate in a group-based diet and physical activity program.
  ACHIEVE: The investigators will test two modules of the adapted video-assisted curriculum format of 45 to 60-minute multipurpose classes, which will include a segment on group weight management (~20-30 minutes) and group exercise (~20-30 minutes). Within each module, the group weight management topic varies by week, and within each week the content of the three weight management groups builds gradually and is purposely repeated. Within each module, the group exercise classes will focus on mild to moderate intensity aerobic exercise using an exercise video. In this pilot study, a trained study interventionist will deliver the ACHIEVE-D curriculum.
Period: Overall Study
Arm/Group | Consumers With SMI
Started | 17
Completed | 16
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants With Serious Mental Illness: Consumers with serious mental illness who attend a psychiatric rehabilitation program
Arm/Group | Participants With Serious Mental Illness
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 37.9 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Participants With Serious Mental Illness Satisfaction With ACHIEVE Curriculum as Assessed by a Yes Response to Two Questions
Description: Two questions during focus group:
  * Would want to continue with the ACHIEVE Program (Yes/No)
  * Would recommend the ACHIEVE program to other clients who want to lose weight (Yes/No)
Time Frame: One week post-intervention
Population: 3 participants did not respond
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Serious Mental Illness: Consumers with serious mental illness who attend a psychiatric rehabilitation program will participate in a pilot test of group-based weight management program modules.
Arm/Group | Participants With Serious Mental Illness
Number analyzed (Participants) | 14
Participants
  Would want to continue with the ACHIEVE Program | 12
  Would recommend the ACHIEVE program to other clients who want to lose weight | 13

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Participants With Serious Mental Illness: Consumers with serious mental illness who attend a psychiatric rehabilitation program (PRP) will participate in a group-based diet and physical activity program.
  ACHIEVE: The investigators will test two modules of the adapted video-assisted curriculum format of 45 to 60-minute multipurpose classes, which will include a segment on group weight management (~20-30 minutes) and group exercise (~20-30 minutes). Within each module, the group weight management topic varies by week, and within each week the content of the three weight management groups builds gradually and is purposely repeated. Within each module, the group exercise classes will focus on mild to moderate intensity aerobic exercise using an exercise video. In this pilot study, a trained study interventionist will deliver the ACHIEVE-D curriculum.
Arm/Group | Participants With Serious Mental Illness
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/92/NCT03999892/Prot_SAP_000.pdf